CLINICAL TRIAL: NCT07140120
Title: LiveSMART: A Sequential, Multiple Assignment Randomized Trial to Prevent Falls in Patients With Cirrhosis - Observational Study
Brief Title: LiveSMART Trial to Prevent Falls in Patients With Cirrhosis - Supplementary Study
Acronym: LiveSMART
Status: Active, not recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Elliot B. Tapper, Associate Professor of Internal Medicine, University of Michigan
Other Study IDs: HUM00225275-B; CER-2021C3-24907 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis, Liver; Portal Hypertension
Keywords: Exercise program; Lactulose; Tai-Chi; Fall prevention; Dietary Protein
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers: Caregivers are a relative, spouse, partner, friend or neighbor who has a significant personal relationship with and provides a broad range of assistance for a patient, including consistent involvement in their medical care.

SUMMARY:
The LIVE-SMART supplementary study will assess social determinants of health (income, education, neighborhood deprivation), financial burden (out-of-pocket costs, productivity loss), financial distress (patient and caregiver-reported outcomes), and financial toxicity (healthcare utilization) among LIVE-SMART participants and their caregivers.

Participants for this supplementary study are participants in the primary study (NCT05794555) and their caregivers.

DETAILED DESCRIPTION:
The supplementary study will augment the primary study the following ways: 1) adding longitudinal questionnaires about financial burden, distress, and toxicity among patients and their caregivers, 2) assessing detailed data and healthcare utilization and associated costs, 3) extending study follow-up by 48 weeks from 24 to 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age or older
* Informal caregiver of a participant enrolled in LIVE-SMART
* English speaking

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers are a relative, spouse, partner, friend or neighbor who has a significant personal relationship with and provides a broad range of assistance for a patient, including consistent involvement in their medical care.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Score for Financial Toxicity - Functional Assessment of Chronic Illness Therapy v2 (COST-FACIT) | Up to 72 weeks
  Financial toxicity will be measured using the COST-FACIT v2 tool, a 12-item, validated self-reported scale validated reflecting experiences of the prior 7-days scored 0-44 (with higher scores indicating more toxicity).

SECONDARY OUTCOMES:
Medications | Up to 72 weeks
  Current medications will be recorded at baseline. Changes and/or additions in medications will be recorded at certain follow-up visits.
Work Productivity and Activity Impairment Questionnaire v2 (WPAI) | Up to 72 weeks
  The WPAI will be used to assess caregivers who report employment, work productivity, absenteeism and presenteeism. Absenteeism is the proportion of work hours lost due to caregiving for someone with cirrhosis subtracted from the total planned work hours in one week before completing the questionnaire. Presenteeism is the proportion of hours worked from the total planned work hours multiplied by the participants impairment in productivity while working (a self-assessed Likert scale from 0 to 10 with 10 indicating complete inability to work). The total work productivity impairment (WPI) is the sum of these two per cent components, ranging from 0 to 100% with 0% indicating no impairment and 100% indicating worst possible impairment. In order to aggregate, productivity loss will be multiplied by the average wage inflated to 2023 dollars.
Out-of-pocket Healthcare Cost Questionnaire (OOP) | Up to 72 weeks
  The OOP questionnaire combines questions from two assessments - Client Service Receipt Inventory (CSRI) and questions pulled from the Healthy Retirement Survey (HRS). Costs will be measured at the household-level using items from the CSRI. Out-of-pocket costs associated with insurance premiums, hospitalizations/ED visits, outpatient surgeries/procedures, clinic visits, skilled nursing facility /rehabilitation stays, prescriptions, dental care, in-home medical care, and any additional medical expenses or healthcare services will be assessed. The cost of hours of caregiving will be calculated by converting the reported hours of informal care provided in the month prior to each interview to a five-year total number of hours. In order to aggregate, replacement costs will be calculated by multiplying the hours by average costs of home health care services inflated to 2023 dollars (e.g., $28/hour).

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Tapper, MD, Principal Investigator — University of Michigan; Marina Serper, MD, MS, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Scott & White Research Institute (BSW), Dallas, Texas

IPD SHARING:
Plan to Share IPD: No